CLINICAL TRIAL: NCT02275390
Title: Effects of a Nurse-led Psycho-education Program for People With First-onset Mental Illness in Psychiatric Outpatient Clinic: A Randomized Controlled Trial (Effects of SPBB for Family Caregivers in Psychosis)
Brief Title: Nurse-led Psycho-education Program for People With First-onset Mental Illness (APN-PEP)
Acronym: APN-PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: United Christian Hospital (Other)
Responsible Party: Principal Investigator, Wai-Tong Chien, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2012100368
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Mental Illness
Keywords: psychosis; self-learning; problem solving; randomized controlled trial; family carer; recent-onset psychosis
MeSH Terms: conditions — Mental Disorders; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Repeated measures, two-arm design
  [SPBB: A repeated-measures, two-arm design with 112 outpatients and their family caregivers]
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blind to the group assignment and intervention undertaken and concealed to the participant list.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse-led Psycho-education [SPBB: Self-learning program] (Experimental): The Nurse-led Psychoeducation Program is comprised of eight 2-hour sessions held at every two weeks (over 4 months). The program consists of five themes: (a) orientation and engaging and understanding of mental health/illness, its related behaviors and community support resources; (b) working collaboratively and empowering and minimizing resistance and challenges using motivational interviewing approach; (c) effective interpersonal and communication skills; (d) strategies in coping with mental illness, sleep hygiene and allaying anxiety; and (e) self-review and evaluation and establishing a realistic plan for future.
  [Note: The participants in the SPBB will complete the self-help and problem-solving manual (5 modules) for caregivers of people with psychotic disorders over 20 weeks, together with an orientation, understanding about psychosis and its care and 4 review sessions.]
  Interventions: Behavioral: Nurse-led Psycho-education (or SPBB: self-learning program); Behavioral: Usual Psychiatric Outpatient Care
- Usual Psychiatric Outpatient Care (Active Comparator): Routine psychiatric outpatient care provided by two psychiatric outpatient clinics under study
  [Note: for SPBB trial, routine psychiatric outpatient care provided by two psychiatric outpatient clinics under study]
  Interventions: Behavioral: Usual Psychiatric Outpatient Care

INTERVENTIONS:
Behavioral: Nurse-led Psycho-education (or SPBB: self-learning program) — The program was modified from the psycho-educational, motivation-driven and emotionally supportive programs developed and previously tested by the research team in Chinese people with different kinds of serious mental illness, mainly including schizophrenia spectrum disorders and mood disorders by Chien and his colleagues in 2012, and adherence therapy for people with psychotic disorders by Gray et al. (2010).
  [Note: SPBB consists of 5 modules (Module 1: Caregiver's well-being; Module 2:Getting the best out of support services; Module 3:Well-being of the person with schizophrenia; Module 4:Dealing with the [psychosocial] effects of the illness; and Module 5: Dealing with [physical and mental health] effects of the illness).]
  Other Names: APN-PEP
  Arms: Nurse-led Psycho-education [SPBB: Self-learning program]
Behavioral: Usual Psychiatric Outpatient Care — These services consisted of medical consultation and treatment by the attending psychiatrist (i.e., around every four weeks), brief education sessions (i.e., 3 or 4 one-hour sessions) on mental illness and treatment received by psychiatric nurses, and advices and referrals for community mental health and social welfare services available and/or family counseling by a psychiatric nurse or medical social worker in each clinic.
  Other Names: UPOC

SUMMARY:
The study aims to test the effectiveness of a nurse-led psycho-education program based on motivational interviewing technique for Chinese patients with first-onset mental illness over a 12-month follow-up. A randomized controlled trial will be conducted with 180 Chinese patients with schizophrenia newly referred to one outpatient clinic in Hong Kong. They will be randomly assigned to either the eight-session nurse-led psycho-education program or usual psychiatric outpatient care (both n=90). The patients' general and mental health, illness insight, self-efficacy, services utilization, and hospitalization rates were measured at recruitment and one week, six months and 12 months post-intervention.

Note: Those who were approached in the clinic and not eligible to participate in this trial will be invited to participate in another controlled trial. The controlled trial tests the effects of a self-help problem-solving based bibliotherapy program (SPBB) for Chinese family caregivers in recent onset psychosis (not more than 1 year onset) at one psychiatric clinic, in comparison to routine outpatient service and family support (control group) for 116 randomly selected family caregivers of outpatients with psychotic disorders over a 6-month follow-up.)

DETAILED DESCRIPTION:
The development of APNs in Hong Kong is in line with nursing development internationally. Since 2001, the Hospital Authority has appointed about 530 nurses as APNs, in whom about 50 are in mental health practice. Five of these psychiatric APNs function independently and interdependently with other health care team members to excel to health educators and care coordinators with fulfilments in health assessment, education and care coordination for clients with noticeable mental health problems, being referred to psychiatric outpatient service. A structured one-to-one psycho-education program has been developed and trial run to provide early psychiatric and psychosocial intervention and support to the clients who have been triaged by the psychiatric nurses in two outpatient clinics in the Kowloon East Cluster as categorised as those who present noticeable mental symptoms but low risks of self-harm or violence. These clients are arranged to have their first psychiatrist consultation in the clinic within two to eight weeks following triage. Prior to the consultation appointment, they are referred to the psychiatric APN in the nurse-led clinic for providing further psychosocial health assessment and early intervention and psychological support. As estimated by the clinic staff, there are 60% of the clients (i.e. 60 cases per month) triaged and classified as such category in the two outpatient clinics.

This study aims to evaluate the effectiveness of the one-to-one, nurse-led psycho-education program provided by the psychiatric APN for those newly referred clients with mental health problems on improving their mental and emotional conditions, quality of life, and satisfaction with service, and on reducing their rates of hospitalization and default follow-up in two psychiatric outpatient clinics (OPD) in Kowloon East region of Hong Kong.

Objectives of the study

1. To investigate the effects of the nurse-led psycho-education program for newly referred clients with mental health problems triaged as Category 2 on improving their mental state, anxiety state, insight and treatment attitude, self-efficacy in life situations, general health, and utilisation of and satisfaction with mental health care services provided over a period of 12 months follow-up; and
2. To investigate the effects of the nurse-led psycho-education program on reducing the clients' rate of hospitalization and default follow-up in the psychiatric OPD over the 12-month follow-up.

[Note: Those are not eligible to participate in this trial will be assessed by an Advanced Practice Nurse to join the randomised controlled trial with repeated measures, parallel-group (2-arm) design will be carried out at one psychiatric clinic. This pilot trial aims to evaluate the effects between the treatment group (i.e., a problem-solving based self-learning program, SPBB) and routine outpatient service (control group) for 116 randomly selected family caregivers of outpatients with recent-onset psychosis over a 6-month follow-up. The study outcomes include the caregivers' burden of care, caregiving experiences, and problem-solving abilities, and the patients' mental state, functioning, and re-hospitalization rates. They will be measured at recruitment, one week, and 6 months following the interventions. Objectives of the study are: 1. To investigate the effects of the SPBB program for family caregivers of recent onset psychosis on improving their caregivers' burden of care, caregiving experiences, and problem-solving abilities, and the patients' mental state, and functioning over a period of 6 months follow-up; and 2. To investigate the effects of the SPBB program on reducing the clients' rate of hospitalization and default follow-ups in the psychiatric outpatient clinic over the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-60 years, able to understand Cantonese/Mandarin;
* having the first-onset of the mental illness (psychotic and mood disorders) within the past six months and new referral or contact with mental healthcare services;
* presenting at least moderate to high levels of psychiatric symptoms (i.e., Brief Psychiatric Rating Scale score of >25 out of 126 and/or Chinese version of the Beck's Depression Inventory-II scores of >10 out of 63); and
* indicating no history and low risk of suicide and self-harm.

Exclusion Criteria:

* receiving other psychosocial interventions organized by the clinics or other healthcare organizations; and
* being classified as the highest priority of psychiatric consultation and treatment (i.e., starting their treatment and care plan with their attending psychiatrist and clinic nurse within one week).

[Note: For SPBB study, the inclusion Criteria of the participants include those who are: Hong Kong Chinese residents, aged 18-64; taking care of and living with a family member primarily diagnosed with one psychotic disorder in the past 12 months psychosis will be recruited; able to read and understand Cantonese/Mandarin; and perceived a moderate to high burden of care (measured by Family Burden Interview Schedule (>20 out of 50 scores). Exclusion criteria of family caregivers include those: received or are receiving another family intervention; are having cognitive impairment or learning disability; and/or presented with a recent personal history of a serious mental illness or medical disease that may adversely affect their ability to participate in the intervention.]

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2012-03-01; Primary Completion 2016-05-31 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Perceived burden of care (Chinese version of Family Burden Interview Schedule) | 6 months after completion of intervention [SPBB study only]
  Caregivers' perceived burden of care will be measured by a Chinese version of the 25-item Family Burden Interview Schedule.
Experience of caregiving (Chinese version of Experience of Caregiving Inventory) | 6 months after completion of intervention [SPBB study only]
  The Chinese version of Experience of Caregiving Inventory is a 66-item self-reporting scale that measures experiences of caregiving to a family member with mental illness based on the transactional model of stress-appraisal-coping.
Brief Psychiatric Rating Scale | 12 months after completion of intervention
  The participants' mental status is assessed and rated on a 7-point Likert scale for each item of the 18-item Brief Psychiatric Rating Scale.

SECONDARY OUTCOMES:
Coping style (42-item Revised Ways of Coping Checklist) | 6 months after completion of intervention [SPBB only]
  A Chinese version of Coping style of the caregivers style will be assessed using the 42-item Revised Ways of Coping Checklist.
Social Problem-Solving (Chinese version of Revised (Short) Social Problem-Solving | 6 months after completion of intervention [SPBB only]
  The Chinese version of Revised (Short) Social Problem-Solving Inventory will be used to assess participants' problem solving.
Mental state (Positive and Negative Syndrome Scale) | 6 months after completion of intervention [SPBB only]
  Patients' mental state will be evaluated by the Positive and Negative Syndrome Scale, a 30-item inventory assessing the absence/severity of psychotic symptoms across positive symptoms, negative symptoms and general psycho-pathology symptoms.
Hospitalization and Default Follow-up Rate | 12 months after completion of intervention [6 months in SPBB study]
  Frequency and length of hospitalizations and outpatient clinic default follow-up rates of participants during intervention and 6 months after interventions would be calculated.
Patient functioning (43-item Specific Level of Functioning Scale) | 6 months after completion of intervention [SPBB only]
  The 43-item Specific Level of Functioning Scale will be used to assess 3 functional domains for patients with schizophrenia spectrum disorders, including physical functioning/personal care (12 items), social functioning (14 items) and community living skills (17 items) on a 5-point Likert scale.
Insight and Treatment Attitudes Questionnaire (APN-PEP) | 12 months after completion of intervention
  The 11-item Insight and Treatment Attitudes Questionnaire was designed to measure patients' awareness of illness and insight into their needs for treatment for schizophrenia (McEvoy et al., 1989). Its items are rated on a 3-point scale (0=no insight; 1=partial insight; 2=good insight). The higher the score, the better is the patient's awareness of and insight into mental health problems, possibility of future illness, and willingness to receive treatments.
World Health Organisation Quality of Life Measure - Brief Version | 12 months after completion of intervention
  The 28-item Chinese version of quality of life scale was modified from the World Health Organization Quality of Life 100-item [WHOQoL-100] questionnaire by the World Health Organization in 1995 and translated and validated by Leung, Tay, Cheng, and Lin (1997). Items are structured in four domains, including physical health, psychological, social relationship, and environment (i.e., 7 items for each subscale). They are rated on a 5-point Likert scale with a high score indicating a better quality of life (total score range 28-140).
Perceived Self-efficacy Scale | 12 months after completion of intervention
  The 10-item Perceived Self-efficacy Scale developed by Jerusalem and Schwarzer in 1992 was translated into Chinese by Zhang and Schwarzer (1995). It is a unidimensional, generic measure of one's competence in the management of challenging and stressful encounters in life situations. ). The items are rated on a 4-point Likert scale (1=absolutely correct to 4=absolutely incorrect), with a total score ranging from 10-40.

CONTACTS AND LOCATIONS:
Overall Officials: WT Chien, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - United Christian Psychiatric OPD, Tai Po, New Territories
  - Kwai Chung Hospital, Kwai Chung, New Terrtories

REFERENCES:
- [Background] Chien WT, Bressington D. A randomized controlled clinical trial of a nurse-led structured psychosocial intervention program for people with first-onset mental illness in psychiatric outpatient clinics. Psychiatry Res. 2015 Sep 30;229(1-2):277-86. doi: 10.1016/j.psychres.2015.07.012. Epub 2015 Jul 10. PMID 26193827
- [Background] McCann TV, Lubman DI, Cotton SM, Murphy B, Crisp K, Catania L, Marck C, Gleeson JF. A randomized controlled trial of bibliotherapy for carers of young people with first-episode psychosis. Schizophr Bull. 2013 Nov;39(6):1307-17. doi: 10.1093/schbul/sbs121. Epub 2012 Nov 20. PMID 23172001
- [Background] Chien WT, Lee IY. The schizophrenia care management program for family caregivers of Chinese patients with schizophrenia. Psychiatr Serv. 2010 Mar;61(3):317-20. doi: 10.1176/ps.2010.61.3.317. PMID 20194413
- [Background] Chien WT, Leung SF, Yeung FK, Wong WK. Current approaches to treatments for schizophrenia spectrum disorders, part II: psychosocial interventions and patient-focused perspectives in psychiatric care. Neuropsychiatr Dis Treat. 2013;9:1463-81. doi: 10.2147/NDT.S49263. Epub 2013 Sep 25. PMID 24109184
- [Background] Chien WT, Leung SF, Chu CS. A nurse-led, needs-based psycho-education intervention for Chinese patients with first-onset mental illness. Contemp Nurse. 2012 Feb;40(2):194-209. doi: 10.5172/conu.2012.40.2.194. PMID 22554213